CLINICAL TRIAL: NCT03573453
Title: Comparison of Continuous Versus Intermittent Enteral Nutrition in Critically Ill Patients. Effect on Energy and Protein Target Achievement, Tolerance and Incidence of Complications. Monocentric Prospective Randomised Study.
Brief Title: Comparison of Continuous Versus Intermittent Enteral Nutrition in Critically Ill Patients.
Acronym: COINN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT0012018
Record Dates: First submitted 2018-04-17; First posted 2018-06-29 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Nutrition Disorders
Keywords: Critical Care; Enteral Nutrition; Ventilator Associated Pneumonia; Gastric Residual Volume
MeSH Terms: conditions — Nutrition Disorders; Pneumonia, Ventilator-Associated | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent (Experimental): enteral nutrition will be administered via enteral feeding pump as 30-60minutes lasting bolus 6 times per day volume of initial bolus will be 80ml. The volume of bolus will be increased gradually according to tolerance, till the estimated target rate will be reached
  Interventions: Other: enteral nutrition
- Continuous (Experimental): enteral nutrition will be administered via enteral feeding pump for at least 16 hours par day initial rate will be 25ml/hour. The rate will be increased gradually according to tolerance, till the estimated target rate will be reached
  Interventions: Other: enteral nutrition

INTERVENTIONS:
Other: enteral nutrition — administration of enteral nutrition

SUMMARY:
The purpose of the study is to compare continuous versus intermittent strategy for enteral nutrition. The study will examine if there is a difference in achieving nutritional delivery goals, tolerance and number of complications of enteral nutrition.

DETAILED DESCRIPTION:
The study will commence following the Approval by The Ethics Research Committee. All patients admitted to our ICU from the 1st of June 2018 to the 31st of May 2019 will be enrolled after fulfilling the inclusion criteria and in the absence of any exclusion criteria. Informed consent will be requested. Enteral nutrition will be administered via nasogastric of orogastric tube. Patients will be randomised in 2 groups. In the group of patients receiving continuous feeding will be enteral nutrition administered via enteral feeding pump for at least 16 hours par day. In the group of patients receiving intermittent feeding will be enteral nutrition administered as 30-60minutes lasting bolus via enteral feeding pump 6 times per day. Following the administration of the bolus the patient will be placed for 30 minutes in semi-upright sitting position. Enteral nutrition requirement and composition will be standardised with the adoption of international guidelines. In 5 subsequent days from the enteral nutrition commencement will be examined if there is a difference in achieving energy and protein targets, tolerance and number of complications of enteral nutrition in between both groups. As achievement of energy and protein targets will be considered at least 80% of calculated values. The tolerance of enteral nutrition will be evaluated by the clinical examination of the abdomen, presence of diarrhoea, vomiting and the gastric residual volume of at least 0,5 liter. As the complications of enteral nutrition will be regarded the aspiration of gastric contents and ventilator associated pneumonia. Nutritional status parameters will be analysed. the length of hospital stay, ICU length of stay and 28-day mortality will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 80 years
* indication of enteral nutrition with nasogastric or orogastric tube
* Nutrition Risk in the Critically Ill (NUTRIC) score ≥5
* Body mass index between 18 - 50
* mechanical ventilation expected for at least 72 hours

Exclusion Criteria:

* upper gastrointestinal tract surgery in previous medical history
* bowel obstruction
* bowel ischemia
* acute pancreatitis
* severe diarrhoea (>1l/24hours)
* gastrointestinal bleeding
* short bowel syndrome
* malabsorption syndrome in previous medical history
* ongoing enteral nutrition on admission to ICU

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-25 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Energy target | 5 days from initiation of enteral nutrition
  Daily assessment of energy intake in critically ill patients with enteral nutrition.Energy target will be achieved if at least 80% of calculated energy intake will be delivered.

SECONDARY OUTCOMES:
Protein target | 5 days from initiation of enteral nutrition
  Daily assessment of protein intake in critically ill patients with enteral nutrition.Protein target will be achieved if at least 80% of calculated protein intake will be delivered.
Tolerance of enteral nutrition | 5 days from initiation of enteral nutrition
  Measurement of the gastric residual volume
Tolerance of enteral nutrition | 5 days from initiation of enteral nutrition
  Incidence of diarrhoea
Tolerance of enteral nutrition | 5 days from initiation of enteral nutrition
  Incidence of vomiting
Complications of enteral nutrition | 5 days from initiation of enteral nutrition
  Incidence of aspiration and ventilator associated pneumonia
Nutritional status | On admission and day 5 from initiation of enteral nutrition
  Blood test : total serum protein test
Nutritional status | On admission and day 5 from initiation of enteral nutrition
  Blood test : albumin test
Nutritional status | On admission and day 5 from initiation of enteral nutrition
  Blood test : prealbumin test

OTHER OUTCOMES:
ICU and hospital length of stay | through study completion, an average of 3 weeks
28-day mortality | 28 days from randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, prof MD PhD, Study Chair — Masaryk University Brno
Locations (1):
- University Hospital Brno and Masaryk University Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hrdy O, Vrbica K, Strazevska E, Suk P, Souckova L, Stepanova R, Sas I, Gal R. Comparison of continuous versus intermittent enteral nutrition in critically ill patients (COINN): study protocol for a randomized comparative effectiveness trial. Trials. 2020 Nov 23;21(1):955. doi: 10.1186/s13063-020-04866-2. PMID 33228772